CLINICAL TRIAL: NCT04713943
Title: Efficacy of >Your< Iron Syrup Supplementation in Children With Iron Deficiency With or Without Mild Microcytic Anemia - a Double-Blind, Placebo-Controlled Multicentric Clinical Study
Brief Title: Efficacy of >Your< Iron Syrup Supplementation in Children With Dietary Iron Deficiency
Acronym: IRON-SI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PharmaLinea Ltd. (Industry)
Collaborators: Clinres Farmacija d.o.o. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: PhL-2017-IRON-SI
Record Dates: First submitted 2021-01-14; First posted 2021-01-19 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Iron-deficiency
Keywords: Iron Supplement; Iron Deficiency; >Your< Iron Syrup
MeSH Terms: conditions — Anemia, Iron-Deficiency; Iron Deficiencies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- >Your< Iron Syrup (Experimental)
  Interventions: Dietary Supplement: >Your< Iron Syrup
- Placebo (Other)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: >Your< Iron Syrup — Once daily dose of >Your< Iron Syrup in the amount of 1 mg/kg body weight of elemental iron for 12 weeks
  Arms: >Your< Iron Syrup
Other: Placebo — Once daily dose of placebo syrup for 12 weeks
  Arms: Placebo

SUMMARY:
The study evaluates the efficacy and safety of >Your< Iron Syrup, a novel iron-containing dietary supplement, in the management of dietary iron deficiency in children. The study is a randomized, double-blind, placebo-controlled intervention conducted in 16 research centers in Slovenia, collectively enrolling 92 eligible children. Eligibility of children for participation in the study will be determined by screening for hemoglobin and ferritin (combined with C-reactive protein) levels in a sample of capillary blood. Eligible children will receive basic dietary advice on how to increase the consumption of dietary iron and will be invited to participate in the study. Enrolled children will be randomized to either >Your< Iron Syrup arm or to placebo arm in a 3:1 ratio, respectively. Changes in body iron stores (ferritin) and in hematological indices as well as occurence of any adverse events will be monitored after 4 and 12 weeks of once-daily supplementation with either >Your< Iron Syrup or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age 9 months to 6 years (inclusive).
* Signed informed consent for screening and for enrollment (parent or legal guardian).
* Iron deficiency with or without mild microcytic anemia not requiring treatment (ferritin ≤20 µg/l and Hb ≥ 100 g/l in a capillary blood sample).

Exclusion Criteria:

* Hb <100 g/l.
* Anemia due to a cause other than iron deficiency.
* Vegan diet.
* Any known concomitant chronic disease (e. g., chronic inflammation, chronic inflammatory bowel disease, malignancy, kidney and/or liver malfunction, lead poisoning).
* Any known allergies to the components of the investigational product.
* Any known medical, physical, or psychological condition that, in the opinion of the investigator, is incompatible with consumption of the investigational product and/or with the conduct of the study.
* Participation in another clinical study less than 1 month before enrollment or current participation in another clinical study.
* Current consumption of iron-containing medicines or dietary supplements.

Ages: 9 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2017-12-22 (Actual); Primary Completion 2020-06-22 (Actual); Study Completion 2020-06-22 (Actual)

PRIMARY OUTCOMES:
The proportion of children having ferritin >20 µg/l | 12 weeks
  Measurement of ferritin in a capillary blood sample (with concomitant measurement of CRP)

SECONDARY OUTCOMES:
The proportion of children having ferritin >20 µg/l | 4 weeks
  Measurement of ferritin in a capillary blood sample (with concomitant measurement of CRP)
Average change in hemoglobin (Hb) | 4 weeks
  Measurements in a capillary blood sample
Average change in Hb | 12 weeks
  Measurement in a capillary blood sample
Average change in hematocrit (HCT) | 4 weeks
  Measurement in a capillary blood sample
Average change in HCT | 12 weeks
  Measurement in a capillary blood sample
Average change in mean corpuscular volume (MCV) | 4 weeks
  Measurement in a capillary blood sample
Average change in MCV | 12 weeks
  Measurement in a capillary blood sample
Average change in mean corpuscular hemoglobin (MCH) | 4 weeks
  Measurement in a capillary blood sample
Average change in MCH | 12 weeks
  Measurement in a capillary blood sample
Average change in mean corpuscular hemoglobin concentration (MCHC) | 4 weeks
  Measurement in a capillary blood sample
Average change in MCHC | 12 weeks
  Measurement in a capillary blood sample
Assessment of safety | 4 weeks
  Collection and assessment of adverse events
Assessment of safety | 12 weeks
  Collection and assessment of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Janez Jazbec, MD, PhD, Principal Investigator — Department of Pediatric Hematology and Oncology, University Medical Centre Ljubljana
Locations (15):
- Slovenia (15):
  - Community Health Center Dr. Julija Polca Kamnik, Kamnik
  - Community Health Center Koper, Koper
  - Private Pediatric Practice Domagoj Puževski, Krško
  - Community Health Center Laško, Laško
  - Community Health Center Ljubljana - Moste-Polje, PE Polje, Ljubljana
  - Community Health Center Ljubljana - Moste-Polje, Ljubljana
  - Community Health Center Ljubljana - PE Rudnik, Ljubljana
  - Community Health Center Ljubljana - Šiška, Ljubljana
  - Department of Pediatric Hematology and Oncology, University Children's Hospital, University Medical Centre Ljubljana, Ljubljana
  - Private Pediatric Practice Ajda Cimperman, Ljubljana
  - Community Health Center dr. Adolf Drolc Maribor, Maribor
  - Community Health Center Medvode, Medvode
  - Private Pediatric Practice Andreja Borinc Beden, Mengeš
  - General Hospital Dr. Franc Derganc Nova Gorica, Šempeter pri Gorici
  - Private Pediatric Practice Pediatrija Šentilj, Šentilj v Slovenskih goricah

IPD SHARING:
Plan to Share IPD: No